CLINICAL TRIAL: NCT00000332
Title: High Dose Nimodipine Pharmacotherapy Adjunct
Brief Title: High Dose Nimodipine Treatment Adjunct - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NIDA-3-0009-1; Y01-3-0009-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Nimodipine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nimodipine

SUMMARY:
The purpose of this study is to determine if nimodipine is more effective than placebo in reducing stimulated craving for cocaine in cocaine dependent individuals denied access to cocaine in inpatient unit.

ELIGIBILITY:
Please contact site for information.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1998-05 (Actual); Primary Completion 2000-01 (Actual); Study Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Stimulated and non-stimulated craving
Stimulated and non-stimulated withdrawal
Anxiety, depression
Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deutsch, M.D., Principal Investigator — Washington D.C. Veterans Affairs Medical Center
Locations (1):
- Washington DC VA, Washington D.C., District of Columbia, United States